CLINICAL TRIAL: NCT07040046
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic, and the Food Effect on the Pharmacokinetics of HS-10542 in Healthy Participants
Brief Title: HS-10542 Study in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10542-101
Record Dates: First submitted 2025-05-08; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: HS-10542; phase 1; Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort1：HS-10542 SAD：HS-10542 capsule (Experimental)
  Interventions: Drug: HS-10542
- Cohort2：HS-10542 Placebo SAD：HS-10542 capsule placebo (Placebo Comparator)
  Interventions: Drug: HS-10542 Placebo
- Cohort3：HS-10542 MAD：HS-10542 capsule (Experimental)
  Interventions: Drug: HS-10542
- Cohort4：HS-10542 Placebo MAD：HS-10542 capsule placebo (Placebo Comparator)
  Interventions: Drug: HS-10542 Placebo

INTERVENTIONS:
Drug: HS-10542 — 1. SAD：HS-10542 capsule (5 predefined dose cohorts ) will be administered orally once on Day 1.
  2. Food Effect [FE] study：HS-10542 capsule (in one predefined dose cohort ) will be administered orally once on Day 15.
  Arms: Cohort1：HS-10542 SAD：HS-10542 capsule
Drug: HS-10542 Placebo — SAD：HS-10542 capsule placebo (5 predefined dose cohorts ) will be administered orally once on Day 1
  Arms: Cohort2：HS-10542 Placebo SAD：HS-10542 capsule placebo
Drug: HS-10542 — MAD：HS-10542 capsule (5 predefined dose cohorts ) will be administered orally once or twice from Day 1 to Day 10.
  Arms: Cohort3：HS-10542 MAD：HS-10542 capsule
Drug: HS-10542 Placebo — MAD：HS-10542 capsule placebo (5 predefined dose cohorts ) will be administered orally once or twice from Day 1 to Day 10.
  Arms: Cohort4：HS-10542 Placebo MAD：HS-10542 capsule placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose escalation phase I clinical study to evaluate the safety, tolerability, pharmacokinetics, and the food effect on the pharmacokinetics of HS-10542 in healthy participants.

DETAILED DESCRIPTION:
This study consists of two parts, of which the Part I consists of the single ascending dose (SAD) study and the food effect (FE) study, while the Part II consists of the multiple ascending dose (MAD) study. The Part I and Part II form this randomized, double-blind, placebo-controlled clinical study to evaluate the safety, tolerability, PK and PD characteristics, as well as the food effect on pharmacokinetics of HS-10542 in Chinese healthy adult participants after single and multiple oral doses.

ELIGIBILITY:
Inclusion Criteria：

1. Male or female between 18 and 64 years of age (critical values inclusive) when signing the informed consent form.
2. Body mass index (BMI = weight/height2) ≥ 19 kg/m2 and ≤ 28 kg/m2 at screening, and body weight ≥ 50 kg for men and ≥ 45 kg for women.
3. Physical examination, laboratory tests, 12-lead ECG, abdominal B-ultrasound and anteroposterior and lateral chest X-ray (or CT) examination showed no abnormality, or slight abnormality but with no clinical significance as judged by the investigator, or slight abnormality but with controllable risk as judged by the investigator, and communication with the sponsor 's medical and pharmacological personnel is required when necessary;
4. Female participants are required to agree to practice highly effective contraception from 2 weeks before screening until 60 days after the last dose:
5. Male participants of childbearing potential are required to agree to practice highly effective contraception from the date of signing the informed consent until 120 days after the last dose; male participants of non-childbearing potential (e.g, having undergone effective sterilization) are required to agree to use additional highly effective contraception in the event of uncertainty about the presence of sperm.
6. Participants should be able to complete vaccinations against Neisseria meningitidis (types A, C, Y, and W-135) and streptococcus pneumoniae at least 2 weeks prior to the first dose, and if participants have previously received the above vaccines, antibody titers or vaccine manufacturer information should be provided, and booster vaccinations should be completed as needed according to local practice guidelines in the opinion of the investigator to obtain adequate protection during the trial.
7. The participants are able to communicate clearly with the investigator, understand and comply with the requirements of this trial, have a comprehensive understanding of the study content, process and possible adverse reactions, and sign the informed consent forms voluntarily.

Exclusion Criteria:

1. Consumed any caffeinated, tea, alcohol, xanthine-rich foods or beverages within 24 hours before administration.
2. Consumed foods known to alter hepatic enzyme activity (eg, pitaya, grapefruit, Seville oranges, etc) and their juice drinks within 1 week before administration.
3. Abnormal vital signs, physical examination, laboratory tests, 12-lead ECG, chest anteroposterior X-ray/CT examination, abdominal ultrasonography, etc. at the time of screening are clinically significant and, as assessed by the investigator, may increase the risk for the participant or affect the interpretation of the study results, which include but are not limited to:

   1. Abnormal liver function: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin (TBiL) ≥ 1.5 times ULN.
   2. Abnormal renal function: eGFR < 60 mL/min/1.73 m2 at screening or abnormal renal function as judged by the investigator, calculated using the estimation formula of Chronic Kidney Disease Epidemiology Collaboration 2021 (CKD-EPI): eGFR (mL/min/1.73 m2) .
   3. Abnormal ECG: The absolute value of QTcF (QT interval corrected by Fridericia 's formula [QT/RR0.33]) > 450 msec for males and > 470 msec for females; or other clinically significant abnormalities as judged by the investigator.
4. Positive hepatitis B virus surface antigen (HBsAg), or negative HBsAg but positive hepatitis B core antibody (HBcAb), or positive HCV Ab, or positive result of any test for HIV antibody or Treponema pallidum-specific antibody at screening and is assessed by the investigator as inappropriate to participate in this trial.
5. participants with inactive, active or latent tuberculosis infection (indicated by tuberculosis on chest X-ray or CT, or positive T-SPOT.TB result) at screening who are assessed as inappropriate for participation in this trial by the investigator.
6. Women with a positive blood pregnancy test result at screening, breastfeeding women, or participants planning to become pregnant during the trial.
7. Used any systemic medication or food (e.g, prescription drugs, over-the-counter drugs, Chinese herbal medicines, health products, special medical supplies, formulas, etc) that could affect the metabolism of investigational drug during the washout period or 5 half-lives (whichever is longer) of a particular drug prior to screening, or participants who are unwilling to undergo washout and discontinue such medication throughout the trial and are assessed as inappropriate for participation in this trial by the investigator. Washout periods for systemic medications or food are detailed in Section 6.7.
8. Those who have been vaccinated with vaccines other than those specified in this protocol within 1 month before screening or are scheduled to be vaccinated within 1 month after the end of the administration.
9. Those who have participated in a clinical trial involving an intervention with another drug or medical device and received an investigational product or use of a medical device within 1 month prior to screening or within 7 half-lives of the other investigational product, whichever is longer.
10. Those who have donated blood or lost blood ≥ 450 mL within 3 months prior to screening, or planning to donate blood during the trial and at the end or within 3 months of the trial.
11. Those who have a known history of smoking (> 5 cigarettes per day on average) within 3 months prior to screening.
12. Those with diseases or medical conditions that may affect the absorption, distribution, metabolism and excretion of oral drugs within 3 months before screening, such as inflammatory bowel disease, peptic ulcer, gastroesophageal reflux disease, chronic diarrhea, subtotal gastrectomy, etc.
13. Those who have a known history of drug abuse/abuse within 6 months prior to screening, or test positive for drug abuse at screening.
14. Those who have a known history of alcohol dependence (an average of ≥ 14 units of alcohol per week, each unit being equivalent to 285 mL of beer, 125 mL of wine, or 25 mL of liquor) within 6 months prior to screening, or a positive breath alcohol test at screening.
15. Those who have undergone ≥ Grade 2 surgery within 6 months before screening, or plan to have surgery or be hospitalized during the trial.
16. Those who have a previous history of severe drug, food or environmental allergy, or known hypersensitivity to the active substance and excipients of the investigational product (including HS-10542 and placebo).
17. Those with a previous history of capsular microorganisms (e.g., meningococcus or pneumococcus) infection, or those with a history of close contact with individuals infected with meningococcal.
18. Those who have difficulty in swallowing solid preparations such as tablets and capsules.
19. Participants who have difficulty in blood collection, and cannot tolerate multiple venous blood draws or have any contraindications to blood collection.
20. Participants with special dietary requirements or inability to comply with the dietary requirements of the study site.
21. As judged by the investigator, those have a history of or currently have any diseases or conditions that may increase the risk of their participation in the trial, affect their compliance with the protocol, or affect their completion of the trial. These include, but are not limited to, diseases or conditions related to the respiratory, circulatory, digestive, urinary, hematological, endocrine, metabolic, nervous, mental, and immune systems.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-12-04 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and the changes in clinical test and examination results | From screening to day 11 or day 21.
  The incidence and severity of adverse events (AEs), serious adverse events (SAEs), and adverse events leading to withdrawal from the study, as well as their correlation with the investigational drug.And the changes in clinical test and examination results before and after administration

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameters：Observed maximum plasma concentration（Cmax） | up to 240 hours after dosing
  The plasma PK parameters to be determined after the first dose in the single ascending dose (SAD) and food effect (FE) studies
Pharmacokinetics (PK) parameters：Time to reach maximum plasma concentration(Tmax） | up to 240 hours after dosing
  The plasma PK parameters to be determined after the first dose in the single ascending dose (SAD) and food effect (FE) studies
Pharmacokinetics (PK) parameters：area under the concentration-time curve from time 0 to time t of last measurable concentration( AUC0-t) | up to 240 hours after dosing
  The plasma PK parameters to be determined after the first dose in the single ascending dose (SAD), food effect (FE), and multiple ascending dose (MAD) studies
PK parameters: Maximum plasma concentration at steady state (Css, max) | up to 240 hours after dosing
  The plasma PK parameters to be determined after the last dose in the MAD study
PK parameters: time to Css, max (Tss, max) | up to 240 hours after dosing
  The plasma PK parameters to be determined after the last dose in the MAD study
PK parameters: Minimum plasma concentration at steady state (Css, min) | up to 240 hours after dosing
  The plasma PK parameters to be determined after the last dose in the MAD study
PK parameters: Area under the plasma concentration-time curve over a dosing interval at steady state (AUCss) | up to 240 hours after dosing
  The plasma PK parameters to be determined after the last dose in the MAD study
PK parameters: Apparent clearance at steady state (CLss/F) | up to 240 hours after dosing
  The plasma PK parameters to be determined after the last dose in the MAD study
PK parameters: Apparent volume of distribution at steady state (Vss/F) | up to 240 hours after dosing
  The plasma PK parameters to be determined after the last dose in the MAD study
PK parameters: Degree of accumulation after multiple doses (Rac) | up to 240 hours after dosing
  The plasma PK parameters to be determined after the last dose in the MAD study
PK parameters: Elimination half-life (t½) | up to 240 hours after dosing
  The plasma PK parameters to be determined after the first dose in the single ascending dose (SAD), food effect (FE), and multiple ascending dose (MAD) studies

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China